CLINICAL TRIAL: NCT06515743
Title: Comparison of Quality of Life After Rehabilitation With an Obturator in Maxillary Defects Due to COVID-19 Associated Mucormycosis and Oral Cancer.
Brief Title: Rehabilitation With an Obturator in Maxillary Defects
Status: Active, not recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, lecturer, Department of Prosthodontics, principle investigator, Menoufia University
Other Study IDs: ADMNF-0020424
Record Dates: First submitted 2024-07-21; First posted 2024-07-23 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Mucormycosis
MeSH Terms: conditions — Mucormycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Delayed surgical obturator — Prosthetic rehabilitation after surgical treatment of mucormycosis is essential for the early restoration of oral function and facial esthetics which is performed by using the surgical obturator.

SUMMARY:
During the COVID-19 pandemic, there was a lot of reporting of COVID-19-associated mucormycosis cases. Managing this condition posed a new challenge to clinicians. Management includes therapeutic drugs and aggressive surgical debridement. Due to the unpredictability of disease prognosis and the possible recurrence of the disease, rehabilitation with delayed surgical obturators is beneficial for patients. Hence, the current study aimed to evaluate the impact of delayed surgical obturators on quality of life of COVID-19-associated mucormycosis patients post-maxillectomies

DETAILED DESCRIPTION:
Globally, the prevalence of mucormycosis varied from 0.005 to 1.7 per million population, while its prevalence is nearly 80 times higher (0.14 per 1000) in India compared to developed countries, in a recent estimate of year 2019-2020.

Among the medical professionals involved in managing patients with mucormycosis, maxillofacial prosthodontists are responsible for prosthetic restoration of lost oral and maxillofacial structures, helping patients to socialize and have an acceptable quality of life after surgical treatment

ELIGIBILITY:
Inclusion Criteria:

*Patients who underwent partial, subtotal and hemi-maxillectomy due to COVID-19-associated mucormycosis and who needed the prosthetic rehabilitation with delayed surgical obturator.

Exclusion Criteria:

* Patients who are unwilling for the study.
* Patients who underwent which bilateral maxillectomies.
* Patients having extensive palatal mucosal loss.

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on 60 patients who underwent maxillectomies between 2020 and 2023. All the patients of 25 years and above who consented for the study were included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Oral healthy related quality of life (oral health impact profile-49)) (OHIP-49) | 6 months
  The OHIP-14 is a self-filled questionnaire developed by Locker and Slade that focuses on 7 dimensions of impact: functional limitation (questions #1,2), physical pain (questions #3,4), psychological discomfort (questions #5,6), physical disability (questions #7,8), psychological disability(question #9,10), social disability (question #11,12), and handicap (question #13,14), with participants being asked to respond according to the frequency of impact on a 5-point Likert scale coded as never (score 0), hardly ever (score 1), occasionally (score2), fairly often (score 3), and very often (score 4). The OHIP-14 is a shorter version of the OHIP-49 but retains the original conceptual dimensions contained in the OHIP-49.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. Elsawy, PhD, Principal Investigator — Menoufia University
Locations (1):
- Mohammed A. El-Sawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD can be shared upon request from the corresponding author.